CLINICAL TRIAL: NCT00828451
Title: Collaborative Research Group for Necrotizing Enterocolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-0105
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Prematurity; Necrotizing Enterocolitis
Keywords: newborn; necrotizing enterocolitis; genetics; growth factors; metabolism
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preterm Infants for EGF Profiles (Experimental): Premature infants born at < 32 weeks gestation who are 7 days old or less. Infants received and intravenous infusion of [5,5,5-2H3]leucine (stable isotope labeled leucine) with sampling of blood, urine and saliva.
  Interventions: Biological: [5,5,5-2H3]leucine (stable isotope labeled leucine)

INTERVENTIONS:
Biological: [5,5,5-2H3]leucine (stable isotope labeled leucine) — intravenous infusion of labeled leucine dissolved in 5% glucose water: priming dose of 18 micromoles (1.8 ml)/kg over 5 minutes, then 18 micromoles (1.8 ml)/hr for 6 hours; one infusion total

SUMMARY:
This proposal will test the hypothesis that synthesis and catabolism of epidermal growth factor (EGF), the genotype of the EGF gene, and the microbiome interact to influence EGF expression in infants at risk for necrotizing enterocolitis (NEC).

DETAILED DESCRIPTION:
* Preterm infants will receive a six hour intravenous infusion of [5,5,5-2H3]leucine (2H3) through an existing intravenous line (IV) to measure EGF synthesis rate.
* Two blood samples will be obtained, one prior to the start of infusion, and one during the infusion. The enrichment of the stable isotope labeled leucine will be measured in the plasma from these samples; DNA will be extracted from the residual cell pellets. The EGF and EGF receptor genes will be sequenced.
* Saliva and urine will be obtained for 5 days following infusion to measure EGF and the rate of incorporation of leucine into EGF using liquid chromatography (LC)/mass spectroscopy (MS)/MS technology, as well as enzyme-linked immunosorbent assay (ELISA) . Saliva will be obtained by a Q tip swab and urine and stool obtained from the diaper.
* Stool will be obtained every 3 to 7 days through 5 weeks to evaluate inflammatory markers and the microbiome.
* If breastfeeding, a single sample of mother's milk will be obtained for measurement of EGF after adequate volumes for infant feeds are achieved.

ELIGIBILITY:
Inclusion Criteria:

* gestation 32 weeks or less
* 1 week of age or less
* intravenous line in place for clinical purposes

Exclusion Criteria:

* imminent death
* active infection
* pre-existing diagnosis of NEC
* fluid or electrolyte imbalance

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hamvas, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Nair RR, Warner BB, Warner BW. Role of epidermal growth factor and other growth factors in the prevention of necrotizing enterocolitis. Semin Perinatol. 2008 Apr;32(2):107-13. doi: 10.1053/j.semperi.2008.01.007. PMID 18346534
- [Background] Warner BB, Ryan AL, Seeger K, Leonard AC, Erwin CR, Warner BW. Ontogeny of salivary epidermal growth factor and necrotizing enterocolitis. J Pediatr. 2007 Apr;150(4):358-63. doi: 10.1016/j.jpeds.2006.11.059. PMID 17382110
- [Background] Spence KL, Zozobrado JC, Patterson BW, Hamvas A. Substrate utilization and kinetics of surfactant metabolism in evolving bronchopulmonary dysplasia. J Pediatr. 2005 Oct;147(4):480-5. doi: 10.1016/j.jpeds.2005.04.039. PMID 16227034
- [Background] Bohlin K, Patterson BW, Spence KL, Merchak A, Zozobrado JC, Zimmermann LJ, Carnielli VP, Hamvas A. Metabolic kinetics of pulmonary surfactant in newborn infants using endogenous stable isotope techniques. J Lipid Res. 2005 Jun;46(6):1257-65. doi: 10.1194/jlr.M400481-JLR200. Epub 2005 Mar 16. PMID 15772427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects admitted to the neonatal intensive care unit at St. Louis Children's Hospital were screened and enrolled from 5/1/2008 to 12/31/2009. Infants born at < 32 weeks and 7 days old or less were eligible for enrollment which occurred in the neonatal intensive care unit or postpartum floor.
Pre-assignment Details: After enrollment 11 of 29 enrolled subjects did not complete the study due to removal of the intravenous line required for infusion, significant deterioration in clinical status resulting in unstable condition as identified by the attending physician, parental withdrawal, and death.
Period: Overall Study
Arm/Group | Preterm Infants for EGF Profiles
Started | 29
Completed | 18
Not Completed | 11
Not completed — Death | 2
Not completed — Lack of intravenous line | 7
Not completed — Withdrawal by Subject | 1
Not completed — Deterioration in clinical status | 1

BASELINE CHARACTERISTICS:
Population: 29 subjects were enrolled. 11 subjects did not complete the study and were not analyzed due to lack of adequate specimens.
Arm/Group | Preterm Infants for EGF Profiles
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Days] | 4 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Salivary EGF (Epidermal Growth Factor) Protein Levels
Description: Salivary EGF protein levels obtained from oral swabs were analyzed by commercially available EGF ELISA kit (R &D systems Inc). EGF protein levels were normalized to micrograms of protein in saliva, and expressed as picogram of EGF protein per microgram of total salivary protein.
Time Frame: Sampling occurred on average day of life 9 with a range from day of life 7 to 21
Population: 29 subjects were enrolled with 11 not completing the study and not analyzed due to lack of specimens
Measure: Median (Full Range); unit: picograms EGF/ microgram of protein
Arm/Group | Preterm Infants for EGF Profiles
Number analyzed (Participants) | 18
picograms EGF/ microgram of protein | 15 [6 to 61]

2. Primary Outcome: Urinary EGF Protein Levels
Description: Urinary EGF protein levels obtained from free flowing urine samples retrieved from subject diaper were analyzed by commercially available EGF ELISA kit (R &D systems Inc). EGF protein levels were normalized to milligrams of creatinine in urine, and expressed as nanograms of EGF protein per milligram of urinary creatinine.
Time Frame: Sampling occurred on average day of life 9 with a range from day of life 7 to 21
Population: 29 subjects were enrolled; 11 did not complete the study and were not analyzed
Measure: Median (Full Range); unit: nanograms of EGF/mg of creatinine
Arm/Group | Preterm Infants for EGF Profiles
Number analyzed (Participants) | 18
nanograms of EGF/mg of creatinine | 48 [7 to 146]

3. Secondary Outcome: EGF Gene Sequencing
Description: Identification of computationally predicted functional variants in EGF gene
Time Frame: Sampling occurred on average day of life 9 with a range from day of life 7 to 21
Population: 29 subjects were enrolled; 11 did not complete the study and were not analyzed
Measure: Number; unit: percentage of participants with variant
Arm/Group | Preterm Infants for EGF Profiles
Number analyzed (Participants) | 18
percentage of participants with variant | 11

ADVERSE EVENTS:
Time Frame: 20 months (5/1/2008 to 12/31/2009)
Groups:
- Preterm Infants for EGF Profile: Premature infants born at < 32 weeks gestation who are 7 days old or less. Infants received and intravenous infusion of [5,5,5-2H3]leucine (stable isotope labeled leucine) with sampling of blood, urine and saliva.
Arm/Group | Preterm Infants for EGF Profile
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
stable isotope labeled EGF could not be detected in the urine and thus the project was closed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No